CLINICAL TRIAL: NCT00502398
Title: Is There Intravascular Hemolysis in Patients With Pulmonary Hypertension?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Other Study IDs: RMC074490CTIL
Record Dates: First submitted 2007-07-15; First posted 2007-07-17 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2007-10

CONDITIONS: Pulmonary Artery Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension | interventions — Hematologic Tests

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood test

SUMMARY:
Patients with hemolytic disorders (e.g. sickle cell anemia or thalassemia) are known to develop pulmonary hypertension. Hemolysis is where red blood cells are destroyed and their contents released into the circulation. It is thought that these red-cell contents cause constriction and thrombosis of the blood vessels in the lungs. Conversely, it is possible that patients with pulmonary hypertension have hemolysis.

In this study we will be drawing blood from a range of patients and normal controls for a panel of blood tests related to hemolysis.

ELIGIBILITY:
Inclusion Criteria:

One of the following four conditions :

* Pulmonary artery hypertension
* Obstructive sleep apnea with pulmonary hypertension
* Lung transplant candidates without pulmonary hypertension
* Normal Controls

Exclusion Criteria:

* Known hemolytic disorder
* Recent blood loss (<3 months)
* Recent blood transfusion (<3 months)
* Liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Kramer, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Pulmonary Institute, Rabin Medical Center (Beilinson campus), Petah Tikva, Israel